CLINICAL TRIAL: NCT00005469
Title: Maturational Changes in Cardiac Structures -- Blood Pressure Relationship -- SCOR in Hypertension
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4914; P50HL044546 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To examine a school-based population of children for maturational changes in blood pressure and cardiac structures.

DETAILED DESCRIPTION:
BACKGROUND:

Although excessive left ventricular mass has been viewed as an adaptation to increased blood pressure, it can precede the rise in blood pressure in hypertensive models. Excessive growth of the heart may reflect additional factors contributing to eventual level of blood pressure. In children, rapid heart growth may be predictive of subsequent high childhood blood pressure level and greater incidence of cardiovascular disease in adult relatives. These studies had the potential of defining maturational changes in known risk factors which might help predict future hypertensive disease.

The study was a subproject within a Specialized Center of Research (SCOR) in Hypertension. The Request for Applications for the SCOR was released in October, 1988.

DESIGN NARRATIVE:

A total of 124 prepubertal males and females were followed longitudinally for five years. Yearly examinations defined the stages of sexual maturation. On four occasions each year, subjects were studied for resting and ambulatory blood pressure, echocardiography, anthropometry and activity assessment. Once yearly, each subject had blood drawn for hormone analyses and whole blood viscosity estimate. From these data, growth velocities of the heart and rate of change of blood pressure were determined. These parameters were analyzed to determine if rapid growth of the heart preceded or followed the rise in blood pressure observed during puberty and body size and composition, sexual maturation and hormone changes, and sympathetic activity.

The study was a subproject within a SCOR in Hypertension. Approximately 7 percent of total dollars were awarded for this subproject.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-09; Study Completion 1996-11 (Actual)

REFERENCES:
- [Background] Mahoney LT, Clarke WR, Burns TL, Lauer RM. Childhood predictors of high blood pressure. Am J Hypertens. 1991 Nov;4(11):608S-610S. doi: 10.1093/ajh/4.11s.608s. PMID 1789940
- [Background] Malcolm DD, Burns TL, Mahoney LT, Lauer RM. Factors affecting left ventricular mass in childhood: the Muscatine Study. Pediatrics. 1993 Nov;92(5):703-9. PMID 8414859
- [Background] Lauer RM, Clarke WR, Mahoney LT, Witt J. Childhood predictors for high adult blood pressure. The Muscatine Study. Pediatr Clin North Am. 1993 Feb;40(1):23-40. doi: 10.1016/s0031-3955(16)38478-4. PMID 8417407
- [Background] Janz KF, Mahoney LT. Three-year follow-up of changes in aerobic fitness during puberty: the Muscatine Study. Res Q Exerc Sport. 1997 Mar;68(1):1-9. doi: 10.1080/02701367.1997.10608861. PMID 9094758
- [Background] Mahoney LT, Burns TL, Stanford W, Thompson BH, Witt JD, Rost CA, Lauer RM. Coronary risk factors measured in childhood and young adult life are associated with coronary artery calcification in young adults: the Muscatine Study. J Am Coll Cardiol. 1996 Feb;27(2):277-84. doi: 10.1016/0735-1097(95)00461-0. PMID 8557894
- [Background] Janz KF, Witt J, Mahoney LT. The stability of children's physical activity as measured by accelerometry and self-report. Med Sci Sports Exerc. 1995 Sep;27(9):1326-32. PMID 8531633
- [Background] Janz KF, Burns TL, Mahoney LT. Predictors of left ventricular mass and resting blood pressure in children: the Muscatine Study. Med Sci Sports Exerc. 1995 Jun;27(6):818-25. PMID 7658942